CLINICAL TRIAL: NCT01278459
Title: Can Atorvastatin Improve Vascular Function in Women With a History of Preeclampsia? A Randomised, Double-blinded, Placebo-controlled Crossover Trial of Atorvastatin in Women With a History of Preeclampsia.
Brief Title: Can Atorvastatin Improve Vascular Function in Women With a History of Preeclampsia?
Acronym: PVS3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2008-005759-21
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Pre-Eclampsia
Keywords: endothelial function; cardiovascular
MeSH Terms: conditions — Pre-Eclampsia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atorvastatin first (Experimental): Participants receive 4 week treatment with atorvastatin 20mg/day, followed by 4 week washout, followed by 4 week treatment with placebo.
  Interventions: Drug: Atorvastatin
- Placebo first (Experimental): Participants receive 4 week treatment with placebo, followed by 4 weeks washout, followed by 4 weeks treatment with atorvastatin 20mg/day.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 4 week treatment, 20mg/day taken orally in tablet form

SUMMARY:
The purpose of the study is to test the hypothesis that a short course of atorvastatin can improve vascular function in women with a history of preeclampsia, compared to placebo.

DETAILED DESCRIPTION:
Women with a history of preeclampsia (high blood pressure/protein in the urine during pregnancy) are at increased risk of developing high blood pressure and heart problems in the 10-15 years after their baby is born. At present we do not know how to reduce this risk. Lowering blood pressure and blood lipid (fats) levels are common strategies for primary prevention of cardiovascular problems. However, most women with a history of preeclampsia in the 5-10 years after pregnancy, will have normal blood pressure readings, blood sugar and cholesterol levels.

Atorvastatin, a type of "statin", is widely used in lowering lipids and preventing cardiovascular disease. This drug has beneficial actions other than lipid-lowering, that may also help prevent cardiovascular problems, including improving function in the lining of blood vessels. We know that impairment in blood vessel function is evident in women in the years after a preeclamptic pregnancy and may contribute to the risk of women after preeclampsia going on to develop cardiovascular disease.

We would like to know if giving a short course of atorvastatin to women with a history of preeclampsia improves their blood vessel function. To do this, ex-preeclamptic women will be invited to take either a atorvastatin or placebo ("dummy") tablet daily for 4 weeks, then no tablets for 4 weeks, then "crossover" to receive the alternative tablet (placebo or atorvastatin) daily for 4 weeks. Blood vessel function would be measured using specialised noninvasive scans and taking a blood test at the beginning and end of each treatment period. The study will be jointly run by the Departments of Cardiovascular Medicine and Obstetrics & Gynaecology at the John Radcliffe Hospital, Oxford.

We anticipate this study will provide valuable data to support larger clinical trials to determine whether improving blood vessel function ultimately reduces the risk of developing early-onset cardiovascular disease after preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Diagnosed with preeclampsia during index pregnancy: defined as (1) new onset hypertension (>140/90 mmHg) after 20 weeks gestation and (2) proteinuria (>0.3g protein/24 hours).
* Participants of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 4 weeks after.
* Participants must be willing to undertake urine pregnancy test at the start of each 4 week phase of the study to exclude unintended pregnancy.
* Participants must have clinically acceptable laboratory markers of renal, thyroid and hepatic function at enrolment.
* Able (in the Investigator's opinion) and willing to comply with all study requirements.
* Willing to allow her General Practitioner and consultant, if appropriate, to be notified of participation in the study and results of clinical laboratory tests.

Exclusion Criteria:

Participants must not be

* Pregnant, lactating during the course of the study.
* Planning pregnancy during course of study or in 4 weeks after study completion
* Taking other medication, whether prescribed or over-the-counter, in the four weeks before first study dose and during the study other than for example mild analgesia or hormonal contraception.
* Taking vitamin medications that may interact with atorvastatin (e.g. niacin, Vitamin D)
* Terminally ill or is inappropriate for placebo medication
* Planning to undertake donation of blood during the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Alteration in brachial artery flow-mediated dilatation | After 4 weeks treatment with atorvastatin or placebo

SECONDARY OUTCOMES:
Microvascular endothelial function as measured by laser doppler flowmetry | After 4 weeks treatment with atorvastatin or placebo
Resistance vessel endothelial function as measured by venous occlusion plethysmography | After 4 weeks treatment with atorvastatin or placebo
Indices of arterial stiffness as measured by arterial tonometry and carotid artery distensibility | After 4 weeks treatment with atorvastatin or placebo
Plasma biomarkers of inflammation and endothelial function | After 4 weeks treatment with atorvastatin or placebo
Endothelial glycocalyx as measured by sublingual Microscan | After 4 weeks treatment with atorvastatin or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, PhD MRCP FESC, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford Department of Cardiovascular Medicine, Oxford, United Kingdom